CLINICAL TRIAL: NCT06196047
Title: Ticagrelor Versus Cilostazol in Ischemic Stroke
Brief Title: Ticagrelor Versus Cilostazol in Minor Ischemic Stroke or TIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23098816
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Ischemic Stroke
Keywords: ticagrelor; acute ischemic stroke; cilostazol; Egypt
MeSH Terms: conditions — Ischemic Stroke | interventions — Ticagrelor; Cilostazol

STUDY DESIGN:
Intervention Model Description: We will conduct our randomized controlled trial, which will contain 2 arms; the ticagrelor arm (group A) will receive (a 180 mg loading dose during the first 24 hours of stroke onset, followed by 90 mg b.i.d from the 2nd to the 90th day). The cilostazol arm will receive (a 200 mg loading dose during the first 24 hours of stroke onset, followed by 100mg twice daily from the 2nd day to the 90th day). All the patients in the two groups will receive aspirin at a loading dose of 75 to 300 mg, followed by 75 mg daily for 21 days.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; in a one-to-one ratio, participants were randomly assigned to receive either loading doses of ticagrelor and aspirin or cilostazol and aspirin by a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 900 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 900. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrolment numbers starting from 1, which were mentioned on their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included ticagrelor and aspirin, and Drug B included cilostazol and aspirin. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ticagrelor arm (Active Comparator): the ticagrelor arm will receive (180 mg loading dose during the first 12 hours of stroke onset followed by 90 mg b.i.d from the 2nd to the 90th day) and aspirin at a loading dose of 75 to 300 mg, followed by 75 mg daily for 21 days.
  Interventions: Drug: Ticagrelor 90 MG
- cilostazol arm (Active Comparator): The cilostazol arm will receive (a 200mg loading dose during the first 12 hours of stroke onset, followed by 100mg twice daily from the 2nd day to the 90th day) and aspirin at a loading dose of 75 to 300 mg, followed by 75 mg daily for 21 days.
  Interventions: Drug: Cilostazol 100 MG

INTERVENTIONS:
Drug: Ticagrelor 90 MG — Efficacy and safety of 180 mg loading dose of ticagrelor administered within 24 hours of first-ever ischemic stroke followed by 90 mg bid for 3 months will be assessed through NIHSS, mRS, new ischemic stroke, and possible adverse effects.
  Other Names: group A
  Arms: ticagrelor arm
Drug: Cilostazol 100 MG — Efficacy and safety of 200 mg loading dose of cilostazol administered within 24 hours of first-ever ischemic stroke followed by 100 mg bid for 3 months will be assessed through NIHSS, mRS, new ischemic stroke, and possible adverse effects.
  Other Names: group B
  Arms: cilostazol arm

SUMMARY:
Along with the current clinical trial, the efficacy and safety of ticagrelor and aspirin administered within the first 24 hours of first-ever ischemic stroke compared to cilostazol and aspirin were assessed through NIHSS, mRS, and possible adverse effects.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial between December 2021 and February 2024 after approval of the ethics committee of the faculty of medicine at Kafr el-Sheik University.

The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will be composed of 2 arms ticagrelor arm, which consisted of 450 patients who received 180 mg loading dose followed by 90 mg b.i.d from the 2nd to the 90th day), and the cilostazol arm consisted of 450 patients who received (a 200mg loading dose during the first 24 hours of stroke onset followed by 100mg twice daily from the 2nd day to the 90th day), All the patients in the two groups received open-label aspirin at a loading dose of 75 to 300 mg, followed by 75 mg daily for 21 days.

Study Procedures:

Every patient in our study will undergo:

Clinical workup: History, clinical assessment & NIHSS were recorded on admission, day 7, and the Modified Rankin Scale as a follow-up after one week and 3 months.

Detection of Risk Factors & Profiles:

Echocardiography& TOE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. - Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

Imaging Follow UP Non-contrast CT brain on admission Day 2 MRI: after 2 days of admission, all the patients in this study will have a brain MRI (stroke protocol; T1W, T2W, FLAIR, DWI, T2 Echo Gradient, MRA of all intra-cerebral vessels).

CT brain: Any patient with unexplained clinical deterioration at any time throughout his/her hospital stay will be urgently imaged by CT.

Primary End Point:

The primary efficacy outcome was the rate of new stroke at 90 days, and the primary safety outcome was the rate of drug hemorrhagic complications using the PLATO bleeding definition.

• Secondary End Point: the secondary efficacy outcomes were to evaluate the rates of patients who achieved a significant reduction in NIHSS (decrease of four points or more) at the seventh day or discharge compared to baseline, the rates of a favorable outcome with (mRS = 0-2) after one week and after 90 days in a face-to-face interview in the outpatient clinic, rates of the composite of recurrent stroke, myocardial infarction and death due to vascular events after 90 days of follow-up, while the secondary safety outcome was the rate of treatment-related adverse effects assessed by a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* the investigators included both genders with eligible ages ranging between 18-75 years, with the first-ever presentation with acute minor ischemic stroke or TIA who received antiplatelet treatment within the first 24 hours of the onset of ischemic stroke. Patients are not eligible for rt-PA treatment

Exclusion Criteria:

* Exclusion Criteria: The investigators excluded patients who had not been followed up on for 90 days after enrollment, those with NIHSS > 4, and patients with a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis, history of head trauma with a residual neurological deficit).

We excluded patients who had clinical seizures at the onset of their stroke, as well as those who had symptoms of any major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks, and those who were on warfarin, regular ticagrelor during the week before admission, or chemotherapy within the previous year.

For safety measures and to avoid associated confounders, we excluded patients with active peptic ulcers, GIT surgery, bleeding history within the last year, and those with a history of major surgery within the last three months.

We ruled out of our trial patients who had a known allergy to the study drugs and those with INR > 1.4 or P.T. >18 or blood glucose level < 50 or > 400 mg/DL or blood pressure < 90/60 or > 185/110 mmHg on admission or Platelets < 100,000.

The investigators considered pregnant and lactating patients or those with stroke due to venous thrombosis, those with wake-up stroke and stroke following cardiac arrest or profuse hypotension ineligible for our trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the rate of new stroke in each group | 90 days
  Assessed during the follow-up period through telephone calls twice per week, a face-to-face interview, and suitable brain imaging in the outpatient clinic once per month and continued for three months
Rate of drug-related hemorrhagic complications | 90 days
  the rate of drug hemorrhagic complications which was evaluated using the PLATO bleeding definition which classified hemorrhagic complications into three types as follows: Major bleeding which had one or more of the following criteria: fatal bleeding, intracranial, intrapericardial, bleeding associated with reduction of hemoglobin > 3-5 g/dl, bleeding required transfusion of two to four units whole blood or PRBCs, bleeding produced hypovolemic shock or severe hypotension that required pressor or surgery; Minor bleeding that required medical intervention to stop or treat bleeding: Minimal bleeding: any bleeding that did not require intervention or treatment such as bruising, bleeding gums, oozing from injection sites.

SECONDARY OUTCOMES:
Value of National Institute of Health Stroke Scale (NIHSS) after one week | 7 days
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid in planning post-acute care disposition.
  It ranges from 0 to 42; the lower the score, the better the stroke condition. The improvement will be counted only if there is a decrease in NIHSS score by four points or more within one week of stroke onset.
value of Modified Rankin Scale (mRS) at one week | 7 days
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome. A favorable stroke outcome is considered with mRS value equals to two or less.
value of Modified Rankin Scale (mRS) at three months | 3 months
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome. A favorable stroke outcome is considered with mRS value equals to two or less.
rate of composite recurrent stroke, myocardial infarction, and death due to vascular events | 3 months
  rates of new stroke, TIA, myocardial infarction, or death from vascular events within three months of treatment, the investigators will perform follow-ups of the patient during visits to the outpatient clinic and perform needed investigations such as brain imaging, Electrocardiography, arterial and venous duplex ultrasound imaging.
rate of drug adverse effects | 90 days
  Drug adverse effects: all side effects related to the drugs of our study will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortiz-Garcia J, Gomez CR, Schneck MJ, Biller J. Recent advances in the management of transient ischemic attacks. Fac Rev. 2022 Jul 22;11:19. doi: 10.12703/r/11-19. eCollection 2022. PMID 35949262
- [Result] Toyoda K, Uchiyama S, Yamaguchi T, Easton JD, Kimura K, Hoshino H, Sakai N, Okada Y, Tanaka K, Origasa H, Naritomi H, Houkin K, Yamaguchi K, Isobe M, Minematsu K; CSPS.com Trial Investigators. Dual antiplatelet therapy using cilostazol for secondary prevention in patients with high-risk ischaemic stroke in Japan: a multicentre, open-label, randomised controlled trial. Lancet Neurol. 2019 Jun;18(6):539-548. doi: 10.1016/S1474-4422(19)30148-6. PMID 31122494
- [Result] Toyoda K, Uchiyama S, Hoshino H, Kimura K, Origasa H, Naritomi H, Minematsu K, Yamaguchi T; CSPS.com Study Investigators. Protocol for Cilostazol Stroke Prevention Study for Antiplatelet Combination (CSPS.com): a randomized, open-label, parallel-group trial. Int J Stroke. 2015 Feb;10(2):253-8. doi: 10.1111/ijs.12420. Epub 2014 Dec 8. PMID 25487817
- [Result] Davis KA, Miyares MA, Dietrich E. Dual antiplatelet therapy with clopidogrel and aspirin after ischemic stroke: A review of the evidence. Am J Health Syst Pharm. 2015 Oct 1;72(19):1623-9. doi: 10.2146/ajhp140804. PMID 26386103
- [Result] Kheiri B, Osman M, Abdalla A, Haykal T, Swaid B, Ahmed S, Chahine A, Hassan M, Bachuwa G, Al Qasmi M, Bhatt DL. Clopidogrel and aspirin after ischemic stroke or transient ischemic attack: an updated systematic review and meta-analysis of randomized clinical trials. J Thromb Thrombolysis. 2019 Feb;47(2):233-247. doi: 10.1007/s11239-018-1786-z. PMID 30511260